CLINICAL TRIAL: NCT06885905
Title: Impact of Chronic Pulmonary Aspergillosis (CPA) on Health Status and Well-being
Acronym: CAPSULE
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government); Tayside Medical Science Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 23IC8471
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pulmonary Aspergillosis
Keywords: CPA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To develop and validate a novel disease-specific questionnaire for measuring HRQoL in patients with Chronic Pulmonary Aspergillosis (CPA-HAQ) for use in clinical research, including clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. All patients >/= 18 years old and able to provide informed consent
2. Patients with a diagnosis of chronic pulmonary aspergillosis
3. To speak and understand English
4. Able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with confirmed Chronic Pulmonary Aspergillosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-08-23 (Estimated); Study Completion 2026-04-23 (Estimated)

PRIMARY OUTCOMES:
Impact of Chronic Pulmonary Aspergillosis (CPA) on health status and Well-being. | 30 months
  To develop and validate a novel disease-specific health-related quality of life (HRQoL) measure in chronic pulmonary aspergillosis (CPA): The Chronic Pulmonary Aspergillosis Health Assessment Questionnaire (CPA-HAQ)

SECONDARY OUTCOMES:
Impact of Chronic Pulmonary Aspergillosis (CPA) on health status and Well-being. | 30 months
  Testing the usability of a newly developed CPA-HAQ measure.
Impact of Chronic Pulmonary Aspergillosis (CPA) on health status and Well-being. | 30 months
  Correlating how HRQoL outcomes relate to existing disease prognostic markers.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Ninewells Hospital & Medical School, Dundee
  - Imperial College London, London
  - Manchester NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NHS Health Research Authority — https://www.hra.nhs.uk/planning-and-improving-research/application-summaries/research-summaries/capsule/